CLINICAL TRIAL: NCT05636111
Title: Phase 1b of Lurbinectedin in Combination With Weekly Paclitaxel and Bevacizumab in Platinum-resistant Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0231; NCI-2022-10037 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Bevacizumab; PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Dose Expansion (Experimental): Pariticipants will be assigned to a dose level of combined paclitaxel, bevacizumab, and lurbinectedin
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab; Drug: Lurbinectedin

INTERVENTIONS:
Drug: Paclitaxel — Given by (IV) vein
  Other Names: Taxol
Drug: Bevacizumab — Given by (IV) vein
  Other Names: Avastin™; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Lurbinectedin — Given by (IV) vein

SUMMARY:
To learn if adding lurbinectedin to the combination of paclitaxel and bevacizumab can help to control advanced cancer.

DETAILED DESCRIPTION:
Primary Objectives:

* To identify dose-limiting toxicities (DLTs) and recommended phase 2 dose (RP2D) of the combination of paclitaxel/bevacizumab/lurbinectedin in women with platinum resistant ovarian cancer.
* To assess macrophage counts by image cytometry in women with platinum resistant ovarian cancer treated with weekly paclitaxel/bevacizumab/lurbinectedin.

Secondary Objectives:

* To assess objective response (OR) and duration of response (DOR).
* To assess clinical benefit rate (CBR), defined as proportion of patients with OR or stable disease (SD) > 4 months.
* To estimate progression free survival (PFS) and overall survival (OS) for at least 12 months

Exploratory Objectives:

--To assess differential effects from baseline, within and between patient treatment cohorts, on macrophage and hypoxia markers, CSF1/R and MHCII, plasma biomarker (VEGF, VEGFR, IL6, IL8, FGF, PDGFAA), tumor and macrophage-derived exosomes, resident macrophage populations in tissue pre-enrollment and after induction bevacizumab (CD11b +CD68, CD11b +CD14/CD15/CD33, CD11b +CD11c, MHCII, CD168+, CD4/CD8, NK, Treg) by multicolor tissue cytometry, as well as serial changes in vivo imaging such as tumor size, macrophage-specific imaging, ADC for cellularity, and DCE for vasculature.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be assessed within 28 days of starting study treatment:

1. Ability to provide signed informed consent in accordance with federal, local, and institutional guidelines.
2. Age ≥ 18 years at time of study entry
3. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
4. Histologically confirmed and documented ovarian, fallopian tube or peritoneal carcinoma: Patients with platinum refractory* or platinum resistant** disease are allowed. Prior anti-VEGF targeted therapy (e.g. bevacizumab, VEGF TKI's) is allowed.

   * Platinum refractory is defined as progression during platinum-containing therapy or within 4 weeks of last dose.
   * Platinum resistant is defined as relapse-free interval 1-6 months of a platinum-containing therapy
5. Prior Therapy: Unlimited prior systemic therapies are allowed.
6. ECOG performance status of 0-1 (Appendix A)
7. Adequate normal organ and marrow function as defined below.

   1. Hemoglobin ≥9.0 g/dL.
   2. Absolute neutrophil count (ANC) > 1500/mm3.
   3. Platelet count ≥100 x 109/L
   4. Serum bilirubin ≤1.5 x ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   5. AST (SGOT)/ALT (SGPT) ≤2.5 x ULN unless liver metastases are present, in which case it must be ≤5x ULN.
   6. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
8. Evidence of post-menopausal status or negative urine or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   2. Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose.
   3. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
9. Measurable disease by RECIST v1.1

Exclusion Criteria:

Exclusion criteria will be assessed within 28 days of starting study treatment. Patients meeting any of the following exclusion criteria are not eligible to enroll in this study.

1. Radiation, chemotherapy, or immunotherapy or any other anticancer therapy ≤2 weeks prior to cycle 1 day 1.
2. Use of an anti-cancer treatment drug or investigational drug during the last 28 days or 5 half-lives (whichever is shorter) prior to cycle 1 day 1. A minimum of 10 days between termination of prior treatment and administration of study treatment is required.
3. Patients with known or suspected conditions likely to increase gastrointestinal toxicity, such as inflammatory bowel disease, bowel obstruction, history of bowel obstruction, or overt bowel involvement by tumor.
4. Patients who are pregnant or lactating.
5. Major surgery </= 28 days prior to cycle 1 day 1.
6. Unstable cardiovascular function:

   1. ECG abnormalities requiring treatment, or
   2. congestive heart failure (CHF) of NYHA Class ≥3, or
   3. myocardial infarction (MI) within 3 months.
7. Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; patients with controlled infection or on prophylactic antibiotics are permitted in the study.
8. Any known history or evidence of hepatitis A, B, or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen); Known to be HIV seropositive
9. Grade >2 peripheral neuropathy at baseline (within 14 days prior to cycle 1 day 1).
10. Serious psychiatric or medical conditions that could interfere with treatment;
11. Participation in an investigational anti-cancer study within 3 weeks prior to Cycle 1 Day 1
12. Concurrent therapy with approved or investigational anticancer therapeutic other than steroids.
13. Patients with coagulation problems and active bleeding within 4 weeks prior to C1D1 (peptic ulcer, epistaxis, spontaneous bleeding)
14. Patients with symptomatic brain lesions
15. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
16. History of hemoptysis (1/2 teaspoon of bright red blood per episode) within 1 month of study enrollment for any tumor type.
17. Non-healing wound, ulcer or bone fracture.
18. Known hypersensitivity to lurbinectedin, paclitaxel, bevacizumab or excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org